CLINICAL TRIAL: NCT05662631
Title: Technology-assisted, In-home Remote Patient Monitoring, Telemedicine, and Home-based Health Care for Treatment of Bone Marrow Transplant Patients.
Brief Title: Remote Monitoring and Home-based Health Care for Treatment of Bone Marrow Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Reimagine Care (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 21-5081.cc
Record Dates: First submitted 2022-11-30; First posted 2022-12-22 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2022-12

CONDITIONS: Bone Marrow Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bone Marrow Transplant Participants (Experimental): Study participants will complete an onboarding session into the Oncology at Home care program prior to discharge from the hospital. During the onboarding process, participants will be introduced to the RC care team, confirm understanding of their customized care plan treatment and goals as established by their BMT care provider, will receive an oral thermometer for use during the study, and will complete patient education. Working with the study team and RC RN, participants will receive, affix, activate, and test a wearable RPM device (the BioIntellisense BioSticker) prior to discharge from the BMT unit. As the BioSticker needs to be replaced every 30 days, patients will also receive three additional BioStickers new in packaging for use during months 2 and 3 as well as to have a back-up device in case of malfunction. Patients will return the BioSticker to BioIntelliSense with the postage paid return envelope provided at discharge.
  Interventions: Device: BioIntellisense BioSticker

INTERVENTIONS:
Device: BioIntellisense BioSticker — This study uses the BioIntellisense BioSticker for RPM, in combination with the BioSync mobile app on participants' mobile phones for data transmission, augmented by use of the BioHub as a backup transmission device. RPM monitoring of device data is accomplished through use of the AlertWatch software system.
  BioSticker System TheBioSticker ® System is an FDA-approved remote monitoring wearable device intended for continuous collection of physiological data in home and healthcare settings. This includes heart rate, respiratory rate, skin temperature, estimated body temperature, frequency of severe cough episodes, activity level, sleep duration, body position, degree of incline while sleeping, step count, step symmetry, step strength, and on/off body times and other symptomatic and biometric data. Data are securely transmitted using AES-CTR 128 bit encryption via wireless connection from the device for storage, review, and further analysis.
  Other Names: BioSticker

SUMMARY:
This study is designed to assess the potential for successfully using technology-assisted in-home oncology care, including remote patient monitoring (RPM), telemedicine, and home-based health care services to support improved care management and appropriate referral to treatment for bone marrow transplant (BMT) patients.

DETAILED DESCRIPTION:
Study participants will complete an onboarding session into the Oncology at Home care program prior to discharge from the hospital. During the onboarding process, participants will be introduced to the RC care team, confirm understanding of their customized care plan treatment and goals as established by their BMT care provider, will receive an oral thermometer for use during the study, and will complete patient education. Working with the study team and RC RN, participants will receive, affix, activate, and test a wearable RPM device (the BioIntellisense BioSticker) prior to discharge from the BMT unit. As the BioSticker needs to be replaced every 30 days, patients will also receive three additional BioStickers new in packaging for use during months 2 and 3 as well as to have a back-up device in case of malfunction. Patients will return the BioSticker to BioIntelliSense with the postage paid return envelope provided at discharge.

The BioSticker will report skin temperature data once per hour, along with additional vital sign information (heart rate, respiratory rate, estimated body temperature, frequency of severe cough episodes, activity level, body position, sleep duration, degree of incline while sleeping, step count, step symmetry, step strength, and on/off body times). Participants will be expected to wear the BioSticker 24 hours per day, 7 days per week, and to also track and log their temperature manually with the oral thermometer according to usual care practice at a minimum of twice per day.

RPM data will be monitored 24 hours per day, 7 days per week by Reimagine Care, Inc. Advanced Practice Providers (APPs) from the Reimagine Care, Inc. Virtual Care Center (VCC). During daytime business hours, APPs will monitor in real time from the VCC. After business hours and on weekends, APPs will be on call and will be automatically notified through a mobile device in case of elevated temperature or other alert of interest. APPs on call will keep the notification device with them at all times.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 89 years old
* Bone marrow transplant recipients (allogeneic)
* Determined by care provider to be stable for discharge to home setting for outpatient care according to clinical practice standard operating procedures (SOPs)
* Residing in the Denver metro area for the duration of the study within 45 minutes of the AMC
* Has in-home caregiver support 24/7 (i.e., does not live alone)
* Has reliable telephone and home internet service and stable wireless network
* Patient has agreed to not submerge the BioSticker device in more than 3 feet of water or submerge for longer than 30 minutes at a time.
* Patient owns or possesses, as the primary user with reliable daily access, a mobile device (iOS or Android) capable of running the study's mobile application and accepting the terms and conditions
* Patient is willing to complete a self-check temperature log to comply and be available for the duration of the study
* Has access to reliable transportation to the hospital 24/7

Exclusion Criteria:

Patients will be excluded from study participation if the PI or designated care provider believes study participation would not be in the patient's best interest for clinical reasons.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-10-16 (Actual); Study Completion 2022-10-16 (Actual)

PRIMARY OUTCOMES:
Number of patients without infection | Up to 90 days
  Number of patients managed at home while using device who did not have an infection. This measure is collected for comparison with alerts. The device does not prevent infection.
Number of alerts detected through RPM | Up to 90 days
  Alert frequency is tracked to evaluate device function for feasibility of use in the clinical workflow. Patient treatment is not alert-based and is dependent on independent clinical confirmation. An alert of interest is defined as any of the following:
  * Oral temperature greater than or equal to 100.4 F (38.0 C) for 1 hour or one reading of 101 F (38.33C);
  * Mean skin temperature over 1 hour > 98.5 F (36.9 C) or 2.5 times standard deviation from patient's baseline over 1 hour;
  * Mean heart rate over 1 hour > 120 beats per minute or 30% overpatient's baseline over 1 hour
  * Mean respiratory rate over 1 hour > 24 breaths per minute or 30% over patient's baseline over 1 hour, does not return to baseline following exertion;
  * The "BioIntelliSense Infection-Like AlertSymptoms" alert will also be monitored.
Number of patients with infection, but without need for hospitalization | Up to 90 days
  Number with infection, without hospitalization, while using device, for comparison with alerts.
Number of patients with infection, with need for hospitalization | Up to 90 days
  Number with infection, with hospitalization, while using device, for comparison with alerts.

SECONDARY OUTCOMES:
Patient satisfaction: Functional Assessment of Cancer Therapy-General (FACT-G) | Baseline
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire that measures Health-related quality of life (HRQoL) in cancer patients. Responses to each question are scored on a 5 point likert scale ranging from 0 (Not at all) to 4 (Very much). Possible total scores range from 0-108, with higher scores indicating a better outcome/better QoL.
Transplant Evaluation Rating Scale (TERS) | Baseline
  The Transplant Evaluation Rating Scale (TERS) measures the predicted impact of psychosocial factors on the successful outcome of transplant. The measurement consists of an expert interview, in which the assessor evaluates 10 distinct domains considered relevant to successful adjustment to the transplant, and rates responses from 1-3. These scores are then weighted for relevance to determine a total weighted score. Possible total scores range from 26.5 to 79.5, with higher scores indicating a worse outcome (greater impairment in psychosocial functioning).
Patient satisfaction: Functional Assessment of Cancer Treatment - Blood/Marrow Transplant (FACT-BMT) | Day 30, Day 90
  The Functional Assessment of Cancer Treatment - Blood/Marrow Transplant (FACT-BMT) assesses quality of life in adult cancer patients undergoing blood & bone marrow transplant. The scale includes 5 subscales. The scores of each scale are summed to compute a total score. Possible total scores range from 0-148. Higher scores indicate a better quality of life and a better outcome.

OTHER OUTCOMES:
Cost of service provision | Up to 90 days
  in US dollars.
Days in hospital in first 90 day post-transplant | Up to 90 days
  In days
Length of hospital stay | Up to 90 days
  In days
Number of ICU admissions post-transplant | Up to 90 days
  Number of ICU admissions
Death rates associated with admission for febrile neutropenia | Up to 90 days
  Number of

CONTACTS AND LOCATIONS:
Overall Officials: Glen E Peterson, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No